CLINICAL TRIAL: NCT00000949
Title: A Randomized, Open-Label, Study of the Impact of Two Doses of Subcutaneous Recombinant IL-2 (Proleukin) on Viral Burden and CD4+ Cell Count in Patients With HIV-1 Infection and CD4+ Cell Counts Greater Than or Equal to 300/mm3
Brief Title: A Study to Evaluate the Effects of Giving Proleukin (rIL-2) to HIV-Positive Patients With CD4 Counts Greater Than 300 Cells/mm3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: CPCRA 059; 11615 (Registry Identifier: DAIDS ES Registry ID)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: AIDS-Related Opportunistic Infections; Interleukin-2; Dose-Response Relationship, Drug; Adolescent Behavior; CD4 Lymphocyte Count; RNA, Viral; Quality of Life; Anti-HIV Agents; Viral Load
MeSH Terms: conditions — HIV Infections; AIDS-Related Opportunistic Infections; Adolescent Behavior | interventions — aldesleukin

INTERVENTIONS:
Drug: Aldesleukin

SUMMARY:
The purpose of this study is to examine how rIL-2 affects HIV-positive patients with CD4 counts over 300 cells/mm3 who are on anti-HIV drug therapy. The drug rIL-2 has been shown to increase CD4 cell counts, which help the body fight off HIV.

There is strong evidence that rIL-2 increases CD4 cell counts (cells of the immune system that fight infection). This study examines the effect of 2 different amounts of rIL-2 on CD4 cell count and the amount of HIV in the blood (viral burden).

DETAILED DESCRIPTION:
There is substantial evidence that rIL-2 increases CD4+ cell count. Whether or not rIL-2 delays progression to AIDS and extends survival is currently unknown, such clinical benefits of rIL-2 can only be established in a large, long-term, randomized trial. This study examines the effect of two different rIL-2 doses on HIV viral burden and CD4+ cell count and provides additional information on optimal dosing, safety, and antiviral activity of rIL-2.

Patients are randomized to receive one of two subcutaneous (sc) doses of recombinant rIL-2 or no rIL-2. Those patients who take rIL-2 initially receive three courses of treatment. For this study, a course is defined as eight calendar weeks, including the five-day period of sc rIL-2 administration. Additional courses are given (no more frequently than every 6 weeks) in order to maintain a CD4+ count of at least twice its baseline level or at least 1,000 cells/mm3. Follow-up will continue for all patients until a common closing date of 12 months following enrollment of the last patient.

ELIGIBILITY:
Inclusion Criteria

You may be eligible for this study if you:

* Are HIV-positive.
* Agree to practice abstinence or use effective birth control methods during the study.
* Are on anti-HIV therapy and have a CD4 count of at least 300 cells/mm3.
* Are at least 18 years old.

Exclusion Criteria

You will not be eligible for this study if you:

* Have a history of progressive diseases.
* Have a history of severe autoimmune/inflammatory disease.
* Have Crohn's disease.
* Are taking antiseizure medications or certain other medications.
* Are receiving chemotherapy.
* Are pregnant or breast-feeding.
* Have ever received rIL-2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460
Dates: Study Completion 2000-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald I. Abrams, Study Chair; Norman Markowitz, Study Chair
Locations (15):
- United States (15):
  - Community Consortium / UCSF, San Francisco, California
  - Denver CPCRA / Denver Public Hlth, Denver, Colorado
  - Washington Reg AIDS Prog / Dept of Infect Dis, Washington D.C., District of Columbia
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - AIDS Research Alliance - Chicago, Chicago, Illinois
  - Louisiana Comm AIDS Rsch Prog / Tulane Univ Med, New Orleans, Louisiana
  - Wayne State Univ - WSU/DMC / Univ Hlth Ctr, Detroit, Michigan
  - Henry Ford Hosp, Detroit, Michigan
  - Southern New Jersey AIDS Clinical Trials, Camden, New Jersey
  - North Jersey Community Research Initiative, Newark, New Jersey
  - Partners in Research / New Mexico, Albuquerque, New Mexico
  - Harlem AIDS Treatment Grp / Harlem Hosp Ctr, New York, New York
  - The Research and Education Group, Portland, Oregon
  - Philadelphia FIGHT, Philadelphia, Pennsylvania
  - Richmond AIDS Consortium / Div of Infect Diseases, Richmond, Virginia

REFERENCES:
- [Background] Abrams DI, Bebchuk JD, Denning ET, Davey RT, Fox L, Lane HC, Sampson J, Verheggen R, Zeh D, Markowitz NP; Terry Beirn Community Programs for Clinical Research on AIDS. Randomized, open-label study of the impact of two doses of subcutaneous recombinant interleukin-2 on viral burden in patients with HIV-1 infection and CD4+ cell counts of > or = 300/mm3: CPCRA 059. J Acquir Immune Defic Syndr. 2002 Mar 1;29(3):221-31. doi: 10.1097/00126334-200203010-00002. PMID 11873071